CLINICAL TRIAL: NCT03964857
Title: Blended Oil Beneficial for Blood Lipids Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: JeyaKumar Henry (Other Government)
Collaborators: Wilmar International Limited (Unknown); National University of Singapore (Other); Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor-Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Organization: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018/00861
Record Dates: First submitted 2019-05-15; First posted 2019-05-28 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Refined olive oil (ROO) (Other): Control
  Interventions: Other: Refined olive oil (ROO)
- Blended Oil 1 (Experimental): BO1, propriety blend of cooking oil containing rice bran, flaxseed and sesame oil blended at proportions different from 'Blended Oil 2
  Interventions: Other: Blended Oil 1 (BO1)
- Blended Oil 2 (Experimental): BO2, propriety blend of cooking oil containing rice bran, flaxseed and sesame oil blended at proportions different from 'Blended Oil 1
  Interventions: Other: Blended Oil 2 (BO2)

INTERVENTIONS:
Other: Refined olive oil (ROO) — Consumption of chicken dishes made with ROO for a period of 8 weeks
  Arms: Refined olive oil (ROO)
Other: Blended Oil 1 (BO1) — Consumption of chicken dishes made with BO1 for a period of 8 weeks
  Arms: Blended Oil 1
Other: Blended Oil 2 (BO2) — Consumption of chicken dishes made with BO2 for a period of 8 weeks
  Arms: Blended Oil 2

SUMMARY:
To investigate the effects of two types of oil blends on blood lipid profile, glucose homeostasis, body composition, gut microflora and other markers of cardiometabolic disease risk in Chinese men and women with borderline hyperlipidemia

DETAILED DESCRIPTION:
The primary aims of this study is to evaluate the effects of consumption of two separate blends of cooking oil, containing rice bran, flaxseed and sesame oils, for a period of 8 weeks, on blood total cholesterol, total triglycerides, low-density and high-density lipoprotein cholesterol and metabolism in borderline hyperlipidaemic, 50 to 70 years old, Chinese, male and postmenopausal female, as compared to refined olive oil. The secondary aims of the study is to evaluate the effect of the two separate blends of cooking oil on markers of cardiometabolic diseases risk (including body composition, glucose homeostasis, markers of oxidative stress and chronic inflammation) and changes in gut microbiota composition and function.

ELIGIBILITY:
Inclusion Criteria:

* Male and post-menopausal female,
* Chinese ethnicity
* Age ≥50 and ≤70 years
* LDL cholesterol (measured) ≥3.06 mmol/l and ≤4.51 mmol/l

Exclusion Criteria:

* Body Mass Index (BMI) > 27.5 kg/m2.
* Having allergies / intolerances to the foods in the meal accompaniments of the study
* Having undergone bariatric surgery
* Having fasting glucose ≥7.0 mmol/l
* Having heart, kidney (nephrotic syndrome), blood or thyroid dysfunctions
* History of chronic liver diseases including NAFLD, liver cirrhosis or hepatic fibrosis or having history of HIV, Hep-B or Hep-C virus
* Having prescription medication or Traditional Chinese Medicine or supplements known to affect blood lipid metabolism, in the opinion of the study investigators, in the last two weeks prior to screening
* Having diabetes or chronic gastrointestinal disorders
* Following any special diets (for medical or aesthetic reasons)
* Smoking
* Having had diarrhea in the last 3 months
* Having taken antibiotics in the last 3 months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2024-07-23 (Estimated)

PRIMARY OUTCOMES:
Change from baseline serum total cholesterol | 8 weeks measured every 2 weeks
  Blood will be collected in plain serum tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline serum low density lipoprotein cholesterol | 8 weeks measured every 2 weeks
  Blood will be collected in plain serum tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline serum total high density lipoprotein cholesterol | 8 weeks measured every 2 weeks
  Blood will be collected in plain serum tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline serum total triglycerides | 8 weeks measured every 2 weeks
  Blood will be collected in plain serum tubes after an overnight fast, centrifuged and frozen within 2 hours of collection

SECONDARY OUTCOMES:
Change from baseline of serum glucose | 8 weeks measured every 2 weeks
  Blood will be collected in plain serum tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline of serum insulin | 8 weeks measured every 2 weeks
  Blood will be collected in plain serum tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline in plasma oxidised low density lipoprotein | For 8 weeks measured every 2 weeks
  Blood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collectionBlood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline in plasma fructosamine | 8 weeks measured every 2 weeks
  Blood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collectionBlood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline in plasma glycated albumin | 8 weeks measured every 2 weeks
  Blood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collectionBlood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline in plasma C-reactive protein | 8 weeks measured every 2 weeks
  Blood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collectionBlood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline in plasma Interleukin-6 | 8 weeks measured every 2 weeks
  Blood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collectionBlood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline in plasma Interleukin-1β | 8 weeks measured every 2 weeks
  Blood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collectionBlood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline in plasma Tumor necrosis factor-α | 8 weeks measured every 2 weeks
  Blood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collectionBlood will be collected in EDTA tubes after an overnight fast, centrifuged and frozen within 2 hours of collection
Change from baseline in body fat composition percentage | 8 weeks
  measured using DEXA (Dual-Energy X-ray Absorptiometry)
Change from baseline in bone mineral density | 8 weeks
  measured using DEXA (Dual-Energy X-ray Absorptiometry)
Change from baseline in blood pressure | 8 weeks measured every 2 weeks
  Measured using Omron blood pressure monitor after an overnight fast in a seated posture, at rest. Blood pressure measured for a minimum of 3 times and the average of the final 2 readings were taken, ensuring that they were within 10 mmHg of each other.
Change from baseline in gut microflora composition | 8 weeks measured on days14 and 56
  Assessed using gut metagenome and metatranscriptome profiling
Change from baseline in gut microflora function | 8 weeks measured on days14 and 56
  Assessed using gut metagenome and metatranscriptome profiling
Change from baseline in Body weight | 8 weeks measured every 2 weeks
  Body impedance assessments (BIA)
Change from baseline in segmental % body fat | 8 weeks measured every 2 weeks
  Body impedance assessments (BIA)
Change in body circumference measures | 8 weeks measured every 2 weeks
  Using measuring tape

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haldar S, Ponnalagu S, Osman F, Tay SL, Wong LH, Jiang YR, Leow MKS, Henry CJ. Increased Consumption of Unsaturated Fatty Acids Improves Body Composition in a Hypercholesterolemic Chinese Population. Front Nutr. 2022 Apr 25;9:869351. doi: 10.3389/fnut.2022.869351. eCollection 2022. PMID 35548564
- [Derived] Haldar S, Wong LH, Tay SL, Jacoby JJ, He P, Osman F, Ponnalagu S, Jiang YR, Lian HPR, Henry CJ. Two Blends of Refined Rice Bran, Flaxseed, and Sesame Seed Oils Affect the Blood Lipid Profile of Chinese Adults with Borderline Hypercholesterolemia to a Similar Extent as Refined Olive Oil. J Nutr. 2020 Dec 10;150(12):3141-3151. doi: 10.1093/jn/nxaa274. PMID 33188423